CLINICAL TRIAL: NCT00781677
Title: Using Neuroimaging to Investigate Neurobiological Correlates of Treatment Resistance Associated With Co-morbid Anxiety in Major Depressive Disorder
Brief Title: Using Neuroimaging to Investigate Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Anx_Dep
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorder; Depression; Anxiety
Keywords: Major Depressive Disorder; Depression; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MDD

SUMMARY:
The purpose of this neuroimaging study is to investigate the brain correlates of Major Depressive Disorder with anxiety symptoms as well as potentially identify predictors of treatment outcome.

DETAILED DESCRIPTION:
The purpose of this study is to test whether the structural and functional connectivity between the dorso-lateral prefrontal cortex (DLPFC) and amygdala will decline as symptoms of co-morbid anxiety (Anxiety Factor Score) increase in patients with MDD. This decrease in connectivity will also account for decrease in treatment response. The structural connectivity will be assessed using Diffusion Tensor Imaging (DTI) and the functional connectivity will be assessed using resting state BOLD fMRI.We propose to use the fMRI and DTI to identify biological markers that are associated with treatment response in a cohort of patients with a spectrum of Anxiety Factor Scores.

ELIGIBILITY:
Inclusion Criteria:

* Competent to give informed consent
* Diagnosis of Major Depressive Disorder
* Males and females
* Ages 18-50 years old
* All races and ethnicities
* Able to read, speak, and understand English*

Exclusion Criteria:

* History of psychiatric illness except Major Depressive Disorder, Generalized Anxiety Disorder, Social Phobia, or Specific Phobia
* Alcohol or substance abuse within the last 6 months or alcohol or substance dependence within the last year
* Diagnosis of an organic brain disease
* Serious unstable medical illness
* History of serious head injury
* Unsafe or unable to have an MRI or previous inability to tolerate MRI
* Pregnancy or breast feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10-20 (Actual); Study Completion 2011-01-20 (Actual)

PRIMARY OUTCOMES:
Treatment response-the Quick Inventory of Depressive Symptomatology: Clinician Rated (QIDS-SR) | 8 weeks

SECONDARY OUTCOMES:
Degree of comorbid anxiety-a subset of the Hamilton Rating Scale for Depression will be used to determine the anxiety/somatization factor scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Kozel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States